CLINICAL TRIAL: NCT07361835
Title: Evaluation of the Effectiveness of Using Virtual Reality Glasses in Prehospital Intervention Training for Crush Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, sureyya gumussoy, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-11.1T/50
Record Dates: First submitted 2026-01-12; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Rhabdomyolysis; Virtual Reality; Emergency Medical Services; Disaster Medicine; Crush Injuries
Keywords: Prehospital Care; Paramedics; Simulation Training; Virtual Reality Simulation
MeSH Terms: conditions — Rhabdomyolysis; Crush Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality-based crush syndrome training (Experimental): Participants receive scenario-based three-dimensional virtual reality simulation training for prehospital crush syndrome management using a head-mounted display.
  Interventions: Device: Virtual reality-based crush syndrome training
- Traditional classroom-based theoretical lecture (Active Comparator): Participants receive traditional classroom-based theoretical education for prehospital crush syndrome management.
  Interventions: Other: Traditional theoretical lecture

INTERVENTIONS:
Device: Virtual reality-based crush syndrome training — A scenario-based three-dimensional virtual reality training program focusing on prehospital crush syndrome assessment and management.
  Arms: Virtual reality-based crush syndrome training
Other: Traditional theoretical lecture — Conventional theoretical classroom instruction on prehospital crush syndrome assessment and management.
  Arms: Traditional classroom-based theoretical lecture

SUMMARY:
This research is a randomized controlled study designed to develop and evaluate the effectiveness of a video-based virtual reality (VR) simulation for prehospital intervention training of crush syndrome for paramedic students. The study aims to examine the impact of VR simulation on knowledge levels, satisfaction, and sense of presence among second-year first and emergency aid students at Muğla Sıtkı Koçman University.

DETAILED DESCRIPTION:
The study will be conducted with second-year students enrolled in the first and emergency aid program at Muğla Sıtkı Koçman University, Fethiye Health Services Vocational School. Participants will be assigned to experimental and control groups using simple randomization. The experimental group will receive training via virtual reality (VR) simulation, while the control group will receive traditional theoretical education. Knowledge levels, technology use, satisfaction, and sense of presence will be measured using various validated scales.

ELIGIBILITY:
Inclusion Criteria:

Being a second-year student currently enrolled in the first and emergency aid program at Muğla Sıtkı Koçman University.

Voluntarily providing written informed consent to participate in the study. Having basic technological literacy to use virtual reality equipment.

Exclusion Criteria:

First-year students who have not yet reached the relevant stage of the curriculum.

Students who have previously participated in a similar virtual reality-based crush syndrome simulation.

Students with medical conditions that may be aggravated by VR use (e.g., severe motion sickness, history of seizures).

Refusal to participate voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Prehospital crush syndrome knowledge level | Baseline (pre-test) and immediately after the training session (post-test).
  The knowledge level of participants is measured using the full 'prehospital crush syndrome knowledge level scale'. The scale consists of 32 items covering four sub-dimensions: general knowledge (12 items), treatment (9 items), transport (6 items), and advanced knowledge (5 items). Each correct answer is scored as 1 point, while incorrect or 'no idea' answers are scored as 0. The total score ranges from a minimum of 0 to a maximum of 32. A higher total score indicates a better understanding and a higher knowledge level of prehospital crush syndrome management.

SECONDARY OUTCOMES:
Educational satisfaction level | Immediately after completion of the training intervention.
  Participant satisfaction with the educational method (virtual reality or theoretical lecture) is measured using the 'education method satisfaction form'. This is a single-item numeric rating scale ranging from a minimum of 0 to a maximum of 10. A score of '0' indicates that the participant is not at all satisfied with the teaching method, while higher scores indicate increasing levels of satisfaction, with a score of '10' representing full satisfaction. Higher scores mean a better outcome.
Sense of presence in virtual environment | Immediately after completion of the virtual reality training session
  The sense of presence in the virtual reality environment is measured using the 'presence questionnaire'. This scale assesses various dimensions such as involvement, sensory fidelity, and adaptation. Each item is scored on a 5-point likert scale, ranging from a minimum of 1 to a maximum of 5. For instance, a score of '1' indicates no presence or very poor quality, while a score of '5' indicates a high level of presence or complete naturalness. A higher total score indicates a greater sense of presence and a more immersive virtual reality experience.
Technology usage level | Baseline (pre-test)
  Participants' orientation and interest towards technology are measured using the 'technology usage scale'. This scale consists of 13 items scored on a 5-point likert scale (1 = strongly disagree to 5 = strongly agree). The total score ranges from a minimum of 13 to a maximum of 65. A higher total score indicates a higher level of technology integration, interest, and adaptation to technological innovations in daily life.
Attitude toward virtual reality in education | Immediately after completion of the training session
  Participants' attitudes toward using virtual reality for learning and professional development are measured using the 'virtual reality attitude scale'. The scale consists of 9 items scored on a 5-point likert scale (1 = strongly disagree to 5 = strongly agree). The total score ranges from a minimum of 9 to a maximum of 45. A higher total score indicates a more positive attitude and higher perceived usefulness regarding the integration of virtual reality into educational processes

CONTACTS AND LOCATIONS:
Overall Officials: Süreyya GÜMÜŞSOY, Principal Investigator — Ege University; Süreyya GÜMÜŞSOY, PhD, Principal Investigator — Ege University
Locations (1):
- Muğla Sıtkı Koçman University, Fethiye Health Services Vocational School, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this study (text, tables, figures, and appendices) will be made available to researchers who provide a methodologically sound proposal. The data will be shared to achieve aims in the approved proposal starting 6 months and ending 36 months after publication of the study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting 6 months after publication and will remain accessible for up to 3 years.
Access Criteria: Data requests should be sent via email to the principal investigator.
URL: https://www.mu.edu.tr/tr/personel/aliakgun

REFERENCES:
- [Background] English: Gunduz, F., & Ersoy, G. (2022). Knowledge levels of 112 ambulance service employees regarding field treatment of crush syndrome: Izmir province example. Journal of Prehospital, 7(1), 37-50.
- [Background] English: Panus, U. (2023). Development of an education program to increase the level of knowledge about crush syndrome in paramedic students. Unpublished Master's Thesis, Ege University.
- [Background] Usuda D, Shimozawa S, Takami H, Kako Y, Sakamoto T, Shimazaki J, Inoue J, Nakayama S, Koido Y, Oba J. Crush syndrome: a review for prehospital providers and emergency clinicians. J Transl Med. 2023 Aug 31;21(1):584. doi: 10.1186/s12967-023-04416-9. PMID 37653520
- See also: Medical Subject Headings (MeSH) Home Page. — https://www.nlm.nih.gov/mesh/
- See also: Reports on Crush Syndrome cases after the 2023 Kahramanmaraş Earthquakes. — https://www.bbc.com/turkce/live/64533110?page=16